CLINICAL TRIAL: NCT01694251
Title: Determination of Mitral Valve Area After Mitral Valve Repair Surgery for Mitral Stenosis Using 3-dimensional Transesophageal Echocardiography
Brief Title: Mitral Valve Area Using 3-dimensional Transesophageal Echocardiography
Acronym: MVA
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, professor of Anesthesiology, Konkuk University Medical Center
Other Study IDs: KUH1160027
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Mitral Valve Repair Surgery
Keywords: mitral valve area; pressure half time; 3 dimensional transesophageal echocardiography; computed tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Even during mitral valve repair procedure (MVP) for severe mitral stenosis (MS), the intraoperative assessment of mitral valve area (MVA) is necessary for evaluating the severity of MS before the repair and excluding residual MS for immediate determination of the success of the repair procedure and postoperative prognosis. For this purpose, several methods have been applied by introperative transesophageal echocardiography (TEE): pressure half-time (PHT) of mitral inflow Doppler and 2-dimensional (2D) planimetry methods have been widely used in clinical practice. However, especially after MVP, the PHT method is usually unreliable because it usually underestimates the MVA due to various intraoperative hemodynamic factors.

The authors hypothesized that the MVA determined by 3D TEE would be more accurate than that by PHT during immediate post-MVP procedure in severe MS patients and comparable to postoperative MVA determined by MDCT. Therefore, the present study determined the MVA by using PHT, 3D planimetry and MDCT before and after the MVP procedure in severe MS patients and analyzed them to evaluate 3D TEE's utility for evaluation of MVA.

DETAILED DESCRIPTION:
After obtaining permission of the Institutional Review Board of Konkuk University Medical Center, Seoul, South Korea , patients scheduled to undergo elective MVP due to more than moderate MS and left atrial enlargement with or without atrial fibrillation (AFib) signed written informed consent agreements and prospectively participate in the present study.

In addition to the routine transthoracic echocardiographic evaluation, cardiac CT examination is performed in all recruited patients prior to surgery to determine MVA.

Induction of anesthesia and tracheal intubation are performed after the administration of intravenous etomidate 0.1-0.2 mg/kg and rocuronium 0.9 mg/kg followed by continuous infusion of remifentanil (0.5-1.0 mcg/kg/min). After tracheal intubation, sevoflurane (1.0 inspired vol%) and infusion of rocuronium (0.2 mg/kg/hr) are administered for anesthesia maintenance.

After anesthesia induction, pulmonary artery catheter (PAC) is placed in right internal jugular vein into pulmonary artery by pressure guidance and a 3D TEE probe (X-9™, Philips Medical Systems Andover, MA, USA) is inserted for the comprehensive intraoperative TEE examination using a 3D echocardiographic imaging platform (iE33; Philips Medical Systems, Andover, MA, USA). While momentarily turning off the ventilator, three consecutive velocity-time integrals (VTIs) of mitral inflow Doppler scans were obtained by applying the continuous wave Doppler parallel to the mitral inflow Color Doppler signal in the midesophageal long-axis view. In case of AFib, the biggest VTI among the 5 consecutive VTIs of the mitral inflow Doppler was used for determining PHT to detect maximal mitral inflow among irregular heartbeats. Immediately after recording the VTIs, a live 3D zoom "en face" MV view from the left atrium (LA) or left ventricle (LV) perspective is acquired.

As baseline data, MVA is determined by using PHT method (MVA-PHT): PHT of the mitral inflow deceleration slope is determined using stored mitral inflow Doppler VTI and the MVA are automatically calculated assuming MVA = 220/PHT. At the same time, a 2D image of the smallest MVA perpendicular to the mitral inflow at the maximal MV opening was achieved by post-processing including aligning and cropping of the acquired 3D images with an installed software (3DQ™ in Q-lab™, Philips, USA). MVA was determined by circumferential tracing of the leaflet edges of the MV opening in the cropped and reconstructed tomographic image from stored 3D volume image (MVA-3D) (Fig. 1). All MVA measurements were repeated 3 times within a minimal time interval by the same expert cardiac anesthesiologists with the mean value used for analysis.

All patients got a single type of MVP (Comprehensive Mitral Valve Apparatus Reconstruction™) consisting of following procedures under moderate hypothermic cardiopulmonary bypass (CPB) by one cardiac surgeon: restoration of a sufficient MV opening with repair of anterior or posterior MV leaflets, mitral commissure, and chordate; and lifting posterior annuloplasty using a flexible ready to use band. A Maze operation is additionally performed in patients who associated with Afib.

Immediately after the weaning from the CPB and achieving stable hemodynamics (mean arterial blood pressure > 65 mmHg, heart rate 60-90 beats per minute, cardiac index > 2.0 L/min/m2), MVA-PHT and MVA-3D are determined in the same manner as the baseline data acquisition.

The following intraoperative exclusion criteria are applied: 1) intraoperative conversion to MV replacement due to insufficient repair procedure, 2) the inability to delineate MV opening due to insufficient 3D imaging.

Within 7 postoperative days, the MVA-CT is determined again for comparison to other methods by an expert cardiac radiologist in the same manner which applied preoperatively.

Statistical analyses are conducted using SPSS 18.0 (SPSS Inc., Chicago, IL, USA). To assess intra-observer variability, the MVAs measured by PHT method and 3D planimetry with TEE are analyzed using intraclass correlation coefficient (ICC). The comparisons of MVA-PHT, MVA-3D, and MVA-CT before or after MVP are analysed used a One Way Repeated Measures Analysis of Variance and their pairwise multiple comparisons are performed via the Tukey method. The comparisons of the other continuous variables of echocardiographic findings are performed by paired t or Wilcoxon Signed Rank tests. The linear regression analysis is used to determine possible correlation between MVA by using each method. Data are expressed as mean ± SD (95% confidence interval. CI) or median (25%-75%), and number of the patients. A p value less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo elective mitral valve repair surgery
* more than moderate mitral stenosis
* left atrial enlargement
* signed written informed consent agreements

Exclusion Criteria:

* urgent or emergency case
* other concurrent valvular surgery
* patient age < 18 years,
* reduced left or right ventricular function (ejection fraction < 40%),
* mitral regurgitation grade more than moderate
* repeated surgery for cardiac valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mitral valve repair mitral stenosis
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
mitral valve area determined by 3D planimetry | within 1 hour after the weaning from CPB
mitral valve area determined by pressure-half time | within 1 hour after the weaning from CPB
mital valve area determined by multi-detactor CT scan | within 7 days weaning from CPB

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD PhD, Principal Investigator — Konkuk University
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul, South Korea